CLINICAL TRIAL: NCT05649345
Title: A Single-arm, Open-Label, Dose Escalation , Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of TR64 in Patients With Advanced Solid Tumors
Brief Title: TR64 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tarapeutics Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR64-CN-PI-01
Record Dates: First submitted 2022-11-22; First posted 2022-12-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TR64 (Experimental): Daily doses by oral administration on each day of each 28 day cycle. Starting dose is 25mg, with escalation to 400mg, and subsequent dose escalation using a modified Fibonacci algorithm.
  Interventions: Drug: TR64

INTERVENTIONS:
Drug: TR64 — TR64 tablets will be given daily for 28 days in 28-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons.

SUMMARY:
This is a open-label, dose escalation, accelerated titration combined 3+3 design, phase I study, to evaluate the safety and tolerability, and to determine the RP2D of TR64 when administered qd in patients with advanced solid tumors. Up to 6 cohorts of 1-6 or 3-6 patients each will be treated in the study.

DETAILED DESCRIPTION:
Patients will receive study treatment until criteria for study termination are met. A Safety Follow-up Visit will be conducted 28 days (±7 days) after the last dose of study treatment. Patients who discontinue study treatment for reasons other disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, patient withdraws consent, is lost to follow-up, death, or until the Sponsor stops the study, whichever comes first.

Adverse events will be assessed using the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.

Tumor response will be assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) scan using RECIST 1.1 criteria, assessed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the procedures of the clinical study and participate voluntarily with signed and dated written informed consent form, comply with the requirements of the study protocol.
* Males and/or females at least 18 years old when signing the informed consent form.
* Histologically or cytologically confirmed patients with advanced malignant solid tumors, eligible patients must have failed standard treatment, no standard treatment, or not suitable for standard treatment at this stage as determined by the investigator.
* Measurable disease with at least one lesion amenable to response assessment per RECIST 1.1.
* Eastern cooperative oncology group performance status (ECOG) ≤2 at screening.
* Life expectancy of at least 3 months.
* Acceptable organ function: Absolute neutrophil count(ANC)≥1.5×109/L; Platelet count(PLT)≥90×109/L; Hemoglobin(Hb)≥90 g/L; Total bilirubin(TBIL)≤1.5×Upper limit of normal value(ULN); Alanine aminotransferase(ALT)≤2.5×ULN; Aspartate aminotransferase(AST)≤2.5×ULN; Creatinine clearance ≥50ml/min.
* Fertile male and female must agree to use medically approved contraceptives during the study and within 90 days after the last dose of the study.

Exclusion Criteria:

* Known or suspected allergies to any of the investigational drug composition.
* Medical history and surgical history excluded according to the protocol.
* Any previous medical treatment history exclude from the protocol.
* Abnormal laboratory results exclude from the protocol.
* pregnant and lactating women (currently breast-feeding or less than six months after delivery although not breast-feeding).
* Subjects may not be able to complete the study duo to poor compliance or other reasons, or unsuitable for the study by the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events and Serious Adverse Events | From the first dose to within 28 days after the last dose
  Frequency, duration and severity of Adverse Events and Serious Adverse Events evaluated by NCI CTCAE v5.0
Dose limited toxicities | within 28 days after the first dose
  Incidence of dose limited toxicities
Maximum tolerated dose | Throughout the study for approximately 2 years
  Evaluated by safety review committee
Recommended phaseII dose | Throughout the study for approximately 2 years
  Evaluated by safety review committee

SECONDARY OUTCOMES:
AUClast | within 35 days after the first dose
  Characterize the pharmacokinetic profile of TR64
AUCinf | within 35 days after the first dose
  Characterize the pharmacokinetic profile of TR64
Cmax | within 35 days after the first dose
  Characterize the pharmacokinetic profile of TR64
Tmax | within 35 days after the first dose
  Characterize the pharmacokinetic profile of TR64
CL/F | within 35 days after the first dose
  Characterize the pharmacokinetic profile of TR64
Vz/F | within 35 days after the first dose
  Characterize the pharmacokinetic profile of TR64
Terminal half-life (T1/2) | within 35 days after the first dose
  Characterize the pharmacokinetic profile of TR64

OTHER OUTCOMES:
ORR | Throughout the study for approximately 2 years
  Efficacy-Overall Response Rate
PFS | Throughout the study for approximately 2 years
  Efficacy-Progression Free Survival
DOR | Throughout the study for approximately 2 years
  Efficacy-Duration of Response
CBR | Throughout the study for approximately 2 years
  Efficacy-Clinical Benefit Rate

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, PhD, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Funan Liu, MD, PhD, Principal Investigator — First Hospital of China Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Hospital of China Medical University, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: No